CLINICAL TRIAL: NCT00062738
Title: Treatment of Depression in Patients With Parkinson's Disease
Brief Title: Treatment of Depression in Parkinson's Disease Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 4381
Record Dates: First submitted 2003-06-12; First posted 2003-06-13 (Estimated); Results first posted 2013-03-05 (Estimated); Last update posted 2015-11-24 (Estimated); Status verified 2015-10

CONDITIONS: Parkinson Disease; Depression
Keywords: Parkinson's disease; Parkinson disease; depression; antidepressants; nortriptyline; paroxetine
MeSH Terms: conditions — Parkinson Disease; Depression | interventions — Paroxetine; Nortriptyline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- nortriptyline (Experimental): drug
  Interventions: Drug: Nortriptyline
- paroxetine (Experimental): drug
  Interventions: Drug: paroxetine
- placebo (Placebo Comparator): placebo
  Interventions: Other: placebo

INTERVENTIONS:
Drug: paroxetine — Paroxetine CR 12.5 - 25 mg q hs
  Other Names: Paxil CR
  Arms: paroxetine
Drug: Nortriptyline — nortriptyline 25 - 75 mg q hs
  Other Names: Pamelor
  Arms: nortriptyline
Other: placebo — matching placebo
  Arms: placebo

SUMMARY:
The goal of this study is to evaluate the effectiveness and safety of two antidepressants--nortriptyline and paroxetine, compared to placebo in patients with Parkinson's disease and depression.

DETAILED DESCRIPTION:
Depression is the most common neuropsychiatric disorder found in patients with Parkinson's disease (PD). It causes immense personal suffering and is associated with increased disability and caregiver burden.

Despite the adverse consequences of depression in patients with PD, there are virtually no empirical data to guide clinical treatment. This study will begin to answer some questions on the treatment of depression by testing a SSRI (selective serotonin reuptake inhibitor) antidepressant, paroxetine, a tricyclic antidepressant, nortriptyline, and placebo in a placebo-controlled trial.

A total of 75 patients with PD will be randomized to each of the three arms in a balanced design.

ELIGIBILITY:
inclusion criteria:

* Parkinson's disease without dementia.
* Depression.
* Males or females.

exclusion criteria:

* Psychosis
* Heart block

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2003-06; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Menza, M.D., Principal Investigator — Rutgers, The State University of New Jersey
Locations (1):
- Robert Wood Johnson Medical School, New Brunswick, New Jersey, United States

REFERENCES:
- [Result] Menza M, Dobkin RD, Marin H, Mark MH, Gara M, Buyske S, Bienfait K, Dicke A. A controlled trial of antidepressants in patients with Parkinson disease and depression. Neurology. 2009 Mar 10;72(10):886-92. doi: 10.1212/01.wnl.0000336340.89821.b3. Epub 2008 Dec 17. PMID 19092112
- [Derived] Dobkin RD, Menza M, Bienfait KL, Gara M, Marin H, Mark MH, Dicke A, Friedman J. Depression in Parkinson's disease: symptom improvement and residual symptoms after acute pharmacologic management. Am J Geriatr Psychiatry. 2011 Mar;19(3):222-9. doi: 10.1097/JGP.0b013e3181e448f7. PMID 20808132
- [Derived] Dobkin RD, Menza M, Bienfait KL, Gara M, Marin H, Mark MH, Dicke A, Troster A. The impact of antidepressant treatment on cognitive functioning in depressed patients with Parkinson's disease. J Neuropsychiatry Clin Neurosci. 2010 Spring;22(2):188-95. doi: 10.1176/jnp.2010.22.2.188. PMID 20463113

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited between 10/2003 and 7/2007, from the RWJMS movement disorder clinic and advertising to local support groups.
Pre-assignment Details: Patients who met inclusion and not exclusion criteria were enrolled.
Groups:
- Nortriptyline: Dosing was flexible with decisions on dose being made at each visit (or between visits if the patient was having troublesome side effects) based on efficacy and tolerability. Nortriptyline was started at 25mg and could be increased up to 75 mg.
- Paroxetine: Paroxetine CR was started at 12.5 mg and could be increased up to 37.5 mg, based on investigator discretion. .
- Placebo: Placebo was started at 1 pill and could be increased up to three pills, based on investigator discretion.
Period: Overall Study
Arm/Group | Nortriptyline | Paroxetine | Placebo
Started | 17 | 18 | 17
Completed | 17 | 18 | 17
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Paroxetine: Paroxetine CR was started at 12.5 mg and could be increased up to 37.5 mg.
- Placebo: Placebo was started at 1 pill and could be increased up to three pills.
- Total: Total of all reporting groups
Arm/Group | Nortriptyline | Paroxetine | Placebo | Total
Number analyzed (Participants) | 17 | 18 | 17 | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 11 | 31
  >=65 years | 7 | 8 | 6 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.9 (9.3) | 62.8 (8.1) | 61.4 (9.2) | 62.2 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 5 | 9 | 25
  Male | 6 | 13 | 8 | 27
Region of Enrollment [Number; unit: participants]
  United States | 17 | 18 | 17 | 52

OUTCOME MEASURES:

1. Primary Outcome: Hamilton Depression Scale
Description: total score on HDRS (0-54 higher score is worse)
Time Frame: 8 weeks
Population: intent to treat - total patients in the arm
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | Nortriptyline | Paroxetine | Placebo
Number analyzed (Participants) | 17 | 18 | 17
units on a scale | 10.84 (6.2) | 12.45 (6.36) | 15.81 (5.78)

2. Secondary Outcome: Percent Responders
Description: Percent of patients who had a 50% decrease in total HDRS at 8 weeks
Time Frame: 8 weeks
Population: intent to treat
Measure: Number; unit: percent of patients who were responders
Arm/Group | Nortriptyline | Paroxetine | Placebo
Number analyzed (Participants) | 17 | 18 | 17
percent of patients who were responders | 53 | 11 | 24
Statistical Analysis 1: Comparison: Nortriptyline vs Paroxetine vs Placebo; For the responder analysis, an LOCF approach was used in which a clinical response was operationally defined as at least a 50% reduction in the HAM-D score from baseline to 8 weeks. Clinical response was cross-tabulated with treatment and Fisher exact test was used to distinguish differences among these groups; Test type: Superiority or Other; p < .05, Fisher Exact; Odds Ratio (OR) = 3.7, 95% CI 2-sided [0.8 to 15.9]

ADVERSE EVENTS:
Time Frame: All data were collected between 10/2003 and 7/2007. Data were collected on each individual for the eight week trial.
Arm/Group | Nortriptyline | Paroxetine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/17 | 1/18 | 2/17
Other Adverse Events (participants affected / at risk) | 17/17 | 7/18 | 11/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nortriptyline (N=17) | Paroxetine (N=18) | Placebo (N=17)
fainting (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) — patient was hospitalized for fainting
muscle rigidity (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) — increased parkinsonism
delirium (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nortriptyline (N=17) | Paroxetine (N=18) | Placebo (N=17)
constipation (Gastrointestinal disorders) | 6 (6) | 1 (1) | 1 (1)
dry mouth (Gastrointestinal disorders) | 7 (7) | 1 (1) | 0 (0)
insomnia (Nervous system disorders) | 2 (2) | 0 (0) | 4 (4)
fatigue (General disorders) | 0 (0) | 3 (3) | 2 (2)
orthostatic hypotension (Cardiac disorders) | 2 (2) | 2 (2) | 2 (2)
dizziness (Cardiac disorders) | 2 (2) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
This was only an eight week trial with relatively few participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No